CLINICAL TRIAL: NCT03818204
Title: Clinical Trial to Improve the Magnetic Levator Prosthesis (MLP) Including the Development and Testing of a Novel Adjustable Force System
Brief Title: Clinical Trial to Improve the Magnetic Levator Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Kevin Houston, Assistant Professor of Ophthalmology, Massachusetts Eye and Ear Infirmary
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-166H
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Blepharoptosis; Ptosis, Eyelid; Myasthenia Gravis; Stroke; Traumatic Brain Injury
MeSH Terms: conditions — Blepharoptosis; Myasthenia Gravis; Stroke; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: This is a prospective cross-over study with some aims having double-blind methodology. Randomization and masking will be used in aims 1 and 2 experiments. Aim 1: The spectacle magnet will be rotated to 1 of 4 settings in an order which will be counterbalanced using a Latin Square approach. Patient and experimenters will be masked to the actual force setting. Aim 2: 17 participants were randomized to be fitted first with either through thickness or through height polarization of the lid magnets using an online randomizer by a study staff not involved in the data collection or analysis who will keep the code. Every other subject in the sequence will be balanced to receive the alternative order. Counterbalancing is being used because of the small sample size.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masked/blinded clinical staff will apply the lid magnets polarized either through thickness or through height (counterbalanced) to the study subjects. Also, 10 magnets of different sizes will be placed inside a plastic housing in order to prevent bias (participant and clinical staff will not know the actual size of the magnets) and counterbalance to control for order effect.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental Group baseline (No Intervention): Subjects with ptosis had their interpalpebral fissure measured continuously for 1 minute with no device.
- Experimental Group MLP 0 degree orientation (Experimental): Subjects with ptosis had their interpalpebral fissure measured continuously for 1 minute with the MLP set at 0 degrees polarization angle.
  Interventions: Device: Magnetic Levator Prosthesis (MLP)
- Experimental Group MLP 30 Degree Orientation (Experimental): Subjects with ptosis had their interpalpebral fissure measured continuously for 1 minute with the MLP set at 30 degrees polarization angle.
  Interventions: Device: Magnetic Levator Prosthesis (MLP)
- Experimental Group MLP 60 Degree Orientation (Experimental): Subjects with ptosis had their interpalpebral fissure measured continuously for 1 minute with the MLP set at 60 degrees polarization angle.
  Interventions: Device: Magnetic Levator Prosthesis (MLP)
- Experimental Group MLP 90 Degree Orientation (Experimental): Subjects with ptosis had their interpalpebral fissure measured continuously for 1 minute with the MLP set at 90 degrees polarization angle.
  Interventions: Device: Magnetic Levator Prosthesis (MLP)
- Experimental Group MLP 180 Degree Orientation (Experimental): Subjects with ptosis had their interpalpebral fissure measured continuously for 1 minute with the MLP set at 180 degrees polarization angle.
  Interventions: Device: Magnetic Levator Prosthesis (MLP)

INTERVENTIONS:
Device: Magnetic Levator Prosthesis (MLP) — Neodymium magnet embedded in a glasses frame and a polymer embedded (PDMS) micro-magnet array fitted externally to the upper lid with IV 3000 securement film. The IV 3000 is FDA approved for extended wear on the skin. Tegaderm, which is essentially the same adhesive, is even FDA approved as an eye covering (we used Tegaderm in early studies but switched to IV 3000 for its superior ease of handling based on packaging technique).
  Arms: Experimental Group MLP 0 degree orientation; Experimental Group MLP 180 Degree Orientation; Experimental Group MLP 30 Degree Orientation; Experimental Group MLP 60 Degree Orientation; Experimental Group MLP 90 Degree Orientation

SUMMARY:
Blepharoptosis (incomplete opening of the eyelids) occurs because of a disruption in the normal agonist-antagonist neuro-muscular complex balance. An external device could restore eyelid movement. A newer class of permanent magnets made of alloys of neodymium (Nd), iron (Fe) and boron (B) might provide the technology needed to develop a feasible external magnetic device that could restore eyelid movement.

DETAILED DESCRIPTION:
Blepharoptosis (incomplete opening of the eyelids) occurs because of a disruption in the normal agonist-antagonist neuro-muscular complex balance. An external device, if able to generate an appropriately balanced force, could restore eyelid movement by performing the paralyzed function; for example, a ptotic (droopy) eyelid could be opened, and the functioning eyelid closure muscle could overcome the device's force (Conway, 1973; Barmettler et. al, 2014; Houston et. al, 2014). Despite this seemingly straight-forward application, permanent magnets for eyelid movement disorders have not thus far become an available treatment. It is possible that earlier magnetic materials lacked the strength (at sizes which were acceptable to patients) to effectively restore the blink, or methods of implantation or external mounting were not effective. A newer class of permanent magnets made of alloys of neodymium (Nd), iron (Fe) and boron (B) might provide the technology needed to develop a feasible external magnetic device. They generate the strongest static magnetic fields yet possible, (1.3T compared to 0.4T of conventional ferrite magnets) (Cyrot, 2005) with exceptional uniaxial magnetocrystalline anisotropy, which makes them resistive to demagnetization (Chikazumui, 1997). The increased magnetic force at a fraction of the size has led to attempts for other medical applications including implantation for gastroesophageal reflux disease (Ganz, 2013), in dental prosthetics (Uribe, 2006), ocular reconstructive surgery (de Negreiros, 2012), and glaucoma (Paschalis et. al, 2013). Problems with extended external non-surgical adhesion to the skin of the eyelid may be solved with hydrocolloid-based medical adhesives e.g. Tegaderm™ (Chen, 1997), already used for IV catheter securement, wound dressing, and as a protective eye covering (FDA, 1997). This material is extremely thin, transparent, and oxygen permeable with an established safety profile for days to weeks of wear. The hydrophyllic properties (FDA, 1997) may be beneficial to the eyelids, which are often moist. In our prior work we established proof-of-concept data demonstrating safety and efficacy for temporary management ptosis up to 2 hour per day for 2 weeks. Due to the sensitive force distance relationship characteristics of magnetic fields and variable nature of ptosis (often worsens throughout the day) the MLP required frequent readjustment and consistent correction was difficult to achieve. Other challenges included lid redness with longer wear times (in the participants who wore the MLP longer than instructed), incomplete spontaneous blinking, and difficultly with self-application of the magnetic lid array to the eye lid. This study aims to address these challenges. In order to improve the MLP we will determine the range of force in the target severe ptosis population to open the lid and where blinking is inhibited, determine the best polarity combination between the lid magnets and the spectacle magnet, determine if rotating the spectacle magnet is a good method to allow simple force adjustment via a dial on the side of the frame, determine if custom made frames improve stability of the frame, and create an applicator tool to help participants apply the lid magnet themselves.

ELIGIBILITY:
Inclusion Criteria:

* Experimental:
* Presence of ptosis for at least one eye which obscures the visual axis in the resting position (without frontalis drive, lifting with forehead muscles)
* Moderate cognitive function or better defined as greater than or equal to 18 out of 30 on a pre-screening of the Mini-Mental State Exam
* Age 5 or older

Exclusion Criteria:

* Experimental:
* Absence of blepharoptosis or presence of a corneal ulcer.
* Those with a corneal ulcer are at risk for permanent loss of vision and should be managed with proven methods.
* Age less than 5,
* Severe Cognitive impairment defined as MMSE score <18, behaviors consistent with delirium (combinations of disorientation, hallucinations, delusions, and incoherent speech), or lethargy. These individuals must be excluded since participation requires competent self-care, reliable responses and cooperation during fitting of the devices.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Houston, OD, M. Sc., Principal Investigator — UMass Chan Medical School
Locations (1):
- Schepens Eye Research Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1-ABCDE; 2-BCDAE; 3-CDABE; 4-DABCE; 5-DCBAE; 6-CBADE; 7-BADCE; 8-ADCBE; 9-ACDBE; 10-BDACE; 11-CABDE; 12-DBCAE; 13-BACDE; 14-CBDAE; 15-DCABE; 16-ADBCE; 17-BCADE; 18-CDBAE; 19-DACBE: Where A=0 degrees, B=30 degrees, C=60 degrees, and D=90 degrees, and E=180 degrees.
Period: Overall Study
Arm/Group | 1-ABCDE | 2-BCDAE | 3-CDABE | 4-DABCE | 5-DCBAE | 6-CBADE | 7-BADCE | 8-ADCBE | 9-ACDBE | 10-BDACE | 11-CABDE | 12-DBCAE | 13-BACDE | 14-CBDAE | 15-DCABE | 16-ADBCE | 17-BCADE | 18-CDBAE | 19-DACBE
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Could not close eye due to impaired facial nerve. | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We originally planned to enroll normal vision subjects to assist with testing the study set up and flow, but ended up not doing this. The study was a crossover design so normal vision control was not required, scientifically.
Groups:
- Experimental Group: The purpose of the experimental group is to test the intervention. Participants will have their acuity measured (refraction as needed), slit lamp with Nafl & NEI scale, visual functioning questionnaire (VFQ), cognitive assessment (MOCA).The eye lid will be prepped and video recorded.The masked clinical staff will then apply the polarized magnets and perform a number of measurements to ascertain effectiveness of intervention.
  -Intervention - Magnetic Levator Prosthesis (MLP)
- Control/Normal Vision Group: The purpose of the normal vision group is to test the experimental setup prior to enrolling ptosis patients. If the measurements of the normal vision group are found to be non-different to the experimental group, the data will be pooled.
  -Intervention - Magnetic Levator Prosthesis (MLP)
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control/Normal Vision Group | Total
Number analyzed (Participants) | 19 | 0 | 19
Age, Continuous [Median (Full Range); unit: years] — Population: One participant was screened and enrolled twice at different time points but was ultimately removed both times because of an impaired facial nerve. Another participant was removed because of difficulties with communication and a self-inflicted corneal abrasion.
  years
    number analyzed (Participants) | 16 | 0 | 16
    (all) | 51 [6 to 85] |  | 51 [6 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 |  | 9
  Male | 10 |  | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 2 |  | 2
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 16 |  | 16
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Baseline Interpalpebral Fissure [Mean (Standard Deviation); unit: millimeters] | 4.7 (2.0) |  | 4.7 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Interpalpebral Fissure During Eye Opening
Description: Change in interpalpebral fissure (resting open) at 5 different force settings of the rotatable adjustable force system.
Time Frame: 6 minutes, 1 minute for each rotation position.
Measure: Mean (95% Confidence Interval); unit: millimeters
Groups:
- Experimental Group Baseline: Subjects with ptosis not wearing any device.
- Experimental Group MLP 0 Degree Orientation: Subjects with ptosis wearing the MLP with force set at the 0 degree polarization angle.
- Experimental Group MLP 30 Degree Orientation: Subjects with ptosis wearing the MLP with force set at the 30 degree polarization angle.
- Experimental Group MLP 60 Degree Orientation: Subjects with ptosis wearing the MLP with force set at the 60 degree polarization angle.
- Experimental Group MLP 90 Degree Orientation: Subjects with ptosis wearing the MLP with force set at the 90 degree polarization angle.
- Experimental Group MLP 180 Degree Orientation: Subjects with ptosis wearing the MLP with force set at the 180 degree polarization angle.
Arm/Group | Experimental Group Baseline | Experimental Group MLP 0 Degree Orientation | Experimental Group MLP 30 Degree Orientation | Experimental Group MLP 60 Degree Orientation | Experimental Group MLP 90 Degree Orientation | Experimental Group MLP 180 Degree Orientation
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
millimeters | 4.5 [3.8 to 5.3] | 6.9 [6.0 to 7.9] | 6.2 [5.2 to 7.1] | 6.3 [5.8 to 7.1] | 6.4 [5.9 to 7.6] | 7.1 [6.2 to 8.1]
Statistical Analysis 1: Comparison: Experimental Group Baseline vs Experimental Group MLP 0 Degree Orientation vs Experimental Group MLP 30 Degree Orientation vs Experimental Group MLP 60 Degree Orientation vs Experimental Group MLP 90 Degree Orientation vs Experimental Group MLP 180 Degree Orientation; The effect of angular position was modeled using linear mixed-effects (multiple regression) models. The five angles were randomly mapped for the dependent variable interpalpebral fissure. Because there were repeated measurements on each eye and each participant might respond differently to each angular position, participant and angular position within participant-eye were included as random effects; Test type: Other; p >= 0.46, Regression, Linear

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the duration of the approximately 1-hour study visit.
Groups:
- Experimental Group: The purpose of the experimental group is to test the intervention. Participants will have their acuity measured (refraction as needed), slit lamp with Nafl & NEI scale.The eye lid will be prepped and video recorded.The masked clinical staff will then apply the polarized magnets and perform a number of measurements to ascertain effectiveness of intervention.
  -Intervention - Magnetic Levator Prosthesis (MLP) polarization angles 0 to 180 degrees.
Arm/Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT03818204/Prot_SAP_000.pdf